CLINICAL TRIAL: NCT05649085
Title: Evaluation of Single-unit Implant-supported Prostheses Survival Using CoCr Prosthetic Abutments: Prospective Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neodent (Industry)
Responsible Party: Sponsor
Other Study IDs: CS.O.013
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-02

CONDITIONS: Missing Teeth; Prosthesis Survival
Keywords: dental implants; dental prosthesis
MeSH Terms: conditions — Anodontia; Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Cobalt-Chromium (CoCr) prosthetic abutments — Cobalt-Chromium (CoCr) prosthetic abutments in single-unit implant-supported prostheses

SUMMARY:
The aim of the study is to prospectively evaluate the survival of JJGC Cobalt-Chromium (CoCr) prosthetic abutments in single-unit implant-supported prostheses, to confirm the long-term safety and performance of the devices.

DETAILED DESCRIPTION:
The cobalt-chromium prosthetic abutments are designed to be installed between the implant and prosthesis. CoCr abutment coping, CoCr abutment for crown set, block and CARES® are devices with indication for prostheses.

Data from the scientific literature support the safety and intended performance of these abutments. An observational clinical study design was chosen to augment the clinical data derived from the use of these devices in accordance with the IFU (Instruction for Use) in the daily clinical practice setting, as well as to assess the long-term prosthetic survival rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients who had GM dental implants from JJGC installed at the ILAPEO College, between 2018 and 2022
* Patients who are using a healing abutment or cover screw and are able to install single-unit, screwed or cemented prostheses, in the maxilla or mandible, which require abutments with greater transmucosal height (due to reduced interocclusal height and/or bone loss)
* Patients presenting antagonist teeth to the implant region

Exclusion Criteria:

* Patients presenting contraindications according to the IFU (instructions for use)
* Patients who require the installation of more than 3 single-unit prostheses with CoCr abutments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who were previously subjected to the installation of GM dental implants by JJGC, at the ILAPEO College, between 2018 and 2022, who are using a healing abutment or cover screw, will receive treatment for installation of single-unit prostheses, screwed or cemented, in the maxilla or mandible, using CoCr abutments, in digital or conventional flow. Patients will be followed up and evaluated at different times over a 2-year period.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Prosthesis survival arte | 24 months after provisional prosthesis installation
  Evaluation of the survival rate of implant-supported prostheses using CoCr prosthetic abutments.

SECONDARY OUTCOMES:
Implant survival rate | 24 months after provisional prosthesis installation
  Survival rate of implant rehabilitated with prosthesis using CoCr abutments
Implant success rate | 24 months after provisional prosthesis installation
  Success rate of implant rehabilitated with prosthesis using CoCr abutments
Patient satisfaction | 24 months after provisional prosthesis installation
  Patient satisfaction with the treatment
Clinician Satisfaction | 24 months after provisional prosthesis installation
  Surgeon satisfaction after the installation of the prosthesis regarding the devices used
Adverse events | 24 months after provisional prosthesis installation
  • Occurrence of adverse events, device deficiencies and residual risks related to abutments, prostheses, and oral health.
Risk factors | 24 months after provisional prosthesis installation
  Influence of risk factors on observed results

CONTACTS AND LOCATIONS:
Overall Officials: Waleska Caldas, Study Director — Neodent
Locations (1):
- Instituto Latino Americano de Pesquisa e Ensino Odontológico (ILAPEO), Curitiba, Brazil

IPD SHARING:
Plan to Share IPD: No